CLINICAL TRIAL: NCT02791139
Title: Association of Midlife Dietary and Lifestyle Factors on Cardiac Functional Changes in the Elderly
Acronym: CardiacAging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/628/C
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: Ageing
MeSH Terms: interventions — Manometry; Genetic Testing; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood will be stored for genetic tests and development of cell lines to study genetic risks for aging related diseases and cardiovascular disease.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Healthy Volunteers will undergo the following studying procedures: Cardiovascular Magnetic Resonance Imaging (CMRI) Echocardiography Tonometry Genetic Testing (Blood) Hand-Grip Strength Measurement Body Fat Mass Analysis
  Interventions: Other: Cardiovascular Magnetic Resonance Imaging (MRI); Other: Echocardiography; Other: Tonometry; Other: Genetic Testing (Blood); Other: Hand-Grip Strength Measurement; Other: Body Fat Mass Analysis
- Ageing: Ageing cohort will undergo the following studying procedures:
  Cardiovascular Magnetic Resonance Imaging (CMRI) Echocardiography Tonometry Genetic Testing (Blood) Body Fat Mass Analysis
  Interventions: Other: Cardiovascular Magnetic Resonance Imaging (MRI); Other: Echocardiography; Other: Tonometry; Other: Genetic Testing (Blood); Other: Body Fat Mass Analysis

INTERVENTIONS:
Other: Cardiovascular Magnetic Resonance Imaging (MRI) — Cardiovascular MRI uses interaction of the magnetic properties of body tissues with strong magnetic fields to create heart images.
Other: Echocardiography — To measure heart chamber size, heart function, blood vessel size and blood vessel function. These measurements will help us understand the type and severity of heart failure.
Other: Tonometry — Tonometry is a noninvasive method to obtain arterial pressure waveform
Other: Genetic Testing (Blood) — The blood will be stored for genetic tests and development of cell lines to study genetic risks for aging related diseases and cardiovascular disease.
Other: Hand-Grip Strength Measurement — We will measure your hand grip strength using a standard hand dynamometer which is a portable meter that you will use your hands to press on.
  Groups: Control
Other: Body Fat Mass Analysis — Body composition will be analysed by a body composition analyser machine onto which you will have to stand on.

SUMMARY:
The investigators aim to investigate the association of midlife dietary and lifestyle factors on cardiac functional changes in the elderly. The investigators hypothesize that even in those without clinically manifest cardiovascular disease, the extent of underlying abnormalities in cardiovascular structure and function in the elderly would be independently related to midlife dietary and lifestyle factors.

DETAILED DESCRIPTION:
This proposal will investigate how midlife factors in diet and lifestyle affect various aspects of cardiac structure and function related to ageing. The investigators plan to conduct the study among a sub-cohort of 600 participants from the Singapore Chinese Health Study. Comprehensive information on diet and lifestyle factors had been collected at recruitment and updated in two subsequent follow-up interviews. Candidate nutrition-related blood biomarkers such as vitamins D, homocysteine, fatty acids (short, medium and long-chain) and lipids (LDL, HDL, triglycerides) will be analyzed from samples obtained between 1999 and 2004. The investigators will study effects of smoking, alcohol consumption, sleep duration, physical activity and diet on cardiac ageing. The investigators will study overall dietary pattern, intake of specific items such as fatty acids, soy food, coffee and tea beverages, from validated food frequency questionnaires (FFQ), and nutrients from questionnaire information from this cohort previously obtained.

These nutrient and lifestyle factors will be studied individually, and for their joint or interactive effects on cardiac ageing measurements. Quantitative cardiac ageing-related outcome parameters describing cardiac mass, systolic and diastolic function, and vessel distensibility will be examined by cardiac magnetic resonance imaging. Maximum oxygen uptake (VO2 max) will be calculated based on age, gender, waist circumference, resting heart rate, and exercise habits. Body composition will be analysed by a body composition analyser machine onto which subjects stand on.

ELIGIBILITY:
Inclusion Criteria:

* Who were younger than 60 years at recruitment
* Had been interviewed at baseline and at the two follow-up interviews
* Had provided biospecimens for research previously before the age of 65 years (2000-2004)
* Who will be 65 years or older by 2013

Exclusion Criteria:

* Any known history of heart disease or stroke
* Anticipated life expectancy < 1 year
* Unable to provide written informed consent to participate in the study
* Patients with cancer
* Patients with chronic renal disease
* Any metallic implants

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 600 ageing participants randomly chosen from a current pool of about 5290 surviving cohort participants in the Singapore Chinese Health Study will be recruited.
  200 Healthy Volunteers control group
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
First occurrence of cardiovascular event | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Su-Mei Angela Koh, MBBS, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong JJ, Zhang H, Leng S, Gao F, Zhao X, Tan K, Tan RS, Zhong L, Koh AS. Superior aortic strain and ventriculoarterial coupling in older women are moderately correlated with Framingham 10-year risk. Eur Heart J Imaging Methods Pract. 2025 Jun 4;3(1):qyaf075. doi: 10.1093/ehjimp/qyaf075. eCollection 2025 Jan. PMID 40584917
- [Derived] Wang LYT, Lim WS, Tan RS, Teo LLY, Tan SY, Ooi CH, Ong ACW, Kovalik JP, Goh J, Gao F, Koh AS. Frequency, intensity and duration of physical activity is associated with frailty in older adults with cardiac aging. Sci Rep. 2025 May 5;15(1):15679. doi: 10.1038/s41598-025-00657-4. PMID 40325063
- [Derived] Chng ACC, Tan HC, Teo LLY, Tan RS, Ewe SH, Leng S, Zhao XD, Zhong L, Koh WP, Kovalik JP, Gao F, Koh AS. Associations between glycated haemoglobin and multi-modal imaging markers of early cardiac aging. Geroscience. 2025 Apr;47(2):1911-1921. doi: 10.1007/s11357-024-01387-7. Epub 2024 Oct 14. PMID 39397221
- [Derived] Zhang H, Leng S, Gao F, Kovalik JP, Tan RS, Wee HN, Chua KV, Ching J, Zhao X, Allen J, Wu Q, Leiner T, Zhong L, Koh AS. Longitudinal aortic strain, ventriculo-arterial coupling and fatty acid oxidation: novel insights into human cardiovascular aging. Geroscience. 2024 Dec;46(6):5459-5471. doi: 10.1007/s11357-024-01127-x. Epub 2024 Mar 22. PMID 38514519
- [Derived] Tan YH, Lim JP, Lim WS, Gao F, Teo LLY, Ewe SH, Keng BMH, Tan RS, Koh WP, Koh AS. Obesity in Older Adults and Associations with Cardiovascular Structure and Function. Obes Facts. 2022;15(3):336-343. doi: 10.1159/000521729. Epub 2022 Mar 4. PMID 35249039
- [Derived] Kovalik JP, Zhao X, Gao F, Leng S, Chow V, Chew H, Teo LLY, Tan RS, Ewe SH, Tan HC, Wee HN, Lee LS, Ching J, Keng BMH, Koh WP, Zhong L, Koh AS. Amino acid differences between diabetic older adults and non-diabetic older adults and their associations with cardiovascular function. J Mol Cell Cardiol. 2021 Sep;158:63-71. doi: 10.1016/j.yjmcc.2021.05.009. Epub 2021 May 24. PMID 34033835
- [Derived] Koh AS, Velmurugan B, Gao F, Tan RS, Wong JI, Teo LLY, Keng BMH, Chua SJM, Yuan JM, Koh WP, Cheung C. Value of soluble Urokinase plasminogen activator receptor over age as a biomarker of impaired myocardial relaxation. BMC Geriatr. 2017 Nov 28;17(1):275. doi: 10.1186/s12877-017-0668-0. PMID 29179674